CLINICAL TRIAL: NCT04709601
Title: Efficacy and Mechanism of Action of Methenamine Hippurate (Hiprex™) in the Management of Recurrent Urinary Tract Infections in Women
Brief Title: Efficacy and Mechanism of Action of Methenamine Hippurate (Hiprex™) in Women With Recurring Urinary Tract Infections.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because the study investigator is no longer following these patients as part of this study. They are followed as part of SOC as the study investigator's patients.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Philippe Zimmern, Professor of Urology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-0725
Record Dates: First submitted 2020-12-17; First posted 2021-01-14 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — methenamine hippurate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1 - Patients with negative and positive urine culture (Experimental)
  Interventions: Drug: Hiprex

INTERVENTIONS:
Drug: Hiprex — Patients with negative urine culture will be prescribed Hiprex 1 g PO BID x 1 yr and patients with a positive urine culture will be prescribed antibiotics.
  Other Names: Methenanime hippurate

SUMMARY:
The purpose of this study is to measure the concentration of formaldehyde in the urine of women with recurrent urinary tract infections on Hiprex; and then, assuming its urinary presence is confirmed at the proper acid urinary pH, evaluate if such a therapy has favorable effects in decreasing the rate of recurrent urinary tract infections over time.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 50 - 85
3. Have RUTIs (at least 2 UTIs within the past 6 months or 3 within the past year) -

Exclusion Criteria:

1. Being on antibiotics at baseline (i.e. suppressive therapy or antibiotic therapy for urinary or non-urinary infections)
2. Neurogenic bladder condition
3. Using urinary catheters (including Foley catheter, intermittent catheterization, and suprapubic catheter)
4. Uncontrolled diabetes (HbA1c > 9)
5. Chronic renal failure defined as serum creatinine > 1.5 mg/dL
6. History of liver disease
7. Patients from out of town, in whom follow-up will not be possible
8. Pregnancy
9. Allergy to Hiprex
10. Inability to take Hiprex reliably at home, such as having psychosis, dementia, or swallowing disorders
11. Non-English speakers -

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Urinary Tract Infections | 1 year
  It would be measured by counting the positive urine cultures, or UTI-like episodes requiring antibiotic treatment during the 1 year of the study period.

SECONDARY OUTCOMES:
Number of oral anti-biotic usage | 1 year
  Number of oral-antibiotics use to treat symptomatic UTI episodes
Number of hospital re-admissions | 1 year
  Number of hospitalizations due to urosepsis and pyelonephritis
Number of adverse events related to Hiprex | 1 year
  Number of participants who experience adverse events >= Grade 3, as defined by Common Terminology Criteria for Adverse Events by CTCA version 5.0
Urine acidity levels | 1 year
  Urine acidity levels will be measured by urinary pH at each visit.
Number of urinary tract infection episodes | up to 2 years
  Diagnose of UTI will be measured for this outcome
Severity of UTI symptoms as measured by the UTI Symptom Assessment questionnaire | 1 year
  UTI Symptom Assessment questionnaire measures severity of UTI symptoms. Possible score range from 0 to 3 (0= Did not have 1= Mild 2=Moderate, and 3=Severe), higher score indicates higher severity of UTI symptoms
Duration of intervals between UTI episodes | 1 year
  Duration of intervals will be measured between one UTI episode to the next UTI episode

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Zimmern, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT-Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No